CLINICAL TRIAL: NCT03520504
Title: A Phase Ib Study With Dose Expansion Cohort of Proton Craniospinal Irradiation for Leptomeningeal Metastases From Solid Tumors
Brief Title: Study of Proton Radiation to the Brain and Spinal Cord for Patients With Leptomeningeal Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-205
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Leptomeningeal Metastases
Keywords: Proton Radiation; craniospinal irradiation (CSI); 18-205
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Intervention Model Description: Single-arm, prospective trial with 3+3 dose de-escalation and dose expansion cohort.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Proton Radiation (Experimental): Patients will be enrolled to receive 30Gy (RBE) in 3Gy (RBE) or 25Gy (RBE) in 2.5Gy (RBE) fractions course of proton CSI.
  The first 3 patients will be enrolled at dose level 30Gy (RBE) in 3Gy(RBE) fractions. If 1 or fewer patients develop dose-limiting toxicity (DLT), 3 additional patients will be enrolled. If 1 or fewer of the 6 patients experiences a DLT, the trial will proceed to the dose expansion cohort at 30Gy (RBE) . In contrast, if 2 or more patients experience a treatment DLT, 3 patients will be enrolled at dose level 25Gy (RBE) in 2.5Gy(RBE) fractions. If 1 or fewer patients develop a DLT, an additional three patients will be enrolled. If 2 or more patients experience a DLT at 25Gy, the study will be stopped. If 1 or fewer patients develop a DLT in these 6 patients, the trial will proceed to the dose expansion cohort at 25Gy (RBE) and the 6 patients who were treated in Phase Ib will be included in full assessment of safety and efficacy.
  Interventions: Radiation: Proton craniospinal irradiation (CSI)

INTERVENTIONS:
Radiation: Proton craniospinal irradiation (CSI) — Patients will be enrolled to receive 30Gy (RBE) in 3Gy (RBE) or 25Gy (RBE) in 2.5Gy (RBE) fractions course of proton CSI.

SUMMARY:
The purpose of this study is to find the safest and most effective dose for delivering proton beam to the space containing CSF, brain, and spinal cord, in treating leptomeningeal metastases. The researchers think that using proton beam radiation to treat the space containing CSF, brain, and spinal cord, instead of treating only the areas where the metastasized tumor cells are causing symptoms, would improve the treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must either be of non-reproductive potential (i.e. post-menopausal by history: >/= 60 years old and no menses for 1> year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test within 2 weeks prior to starting treatment.
* Patient with solid tumor malignancy with leptomeningeal metastases established radiographically and/or through CSF cytology.
* KPS ≥ 60.
* Age ≥ 10 years.
* For adult patient, the patient is able to provide informed consent. For pediatric patient, a parent is able to provide informed consent.
* Patient at reproductive potential must agree to practice an effective contraceptive method.
* Adequate bone marrow function:

  * Hemoglobin ≥ 8g/dL
  * Absolute neutrophil count ≥500/mm^3
  * Platelet count ≥ 100,000/mm^3

Exclusion Criteria:

* Patient with multiple, serious major neurologic deficits including encephalopathy.
* Patient with extensive systemic disease and without reasonable systemic treatment options.
* Patient who is unable to undergo MRI brain and spine with gadolinium contrast.
* Previous radiotherapy to the intended treatment site that precludes developing a treatment plan that respects normal tissue tolerances.
* Pregnant or lactating women.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
number of patients with dose-limiting toxicity | 2 years
  will be assessed by physician-graded CTCEAv4

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Higginson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm